CLINICAL TRIAL: NCT06752551
Title: Apprehension-based Training Compared With Standard Physical Therapy Among Military Personnel Following Anterior Shoulder Dislocation
Brief Title: Apprehension-based Training Compared With Standard Physical Therapy for Military Personnel Following Anterior Shoulder Dislocation - a Randomized Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alon Rabin (Other)
Collaborators: Medical Corps, Israel Defense Force (Other)
Responsible Party: Sponsor-Investigator, Alon Rabin, Principal investigator, Ariel University
Organization: Ariel University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2388-2023
Record Dates: First submitted 2024-12-22; First posted 2024-12-30 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Anterior Shoulder Dislocation
Keywords: Randomized clinical trial; Anterior shoulder dislocation; Shoulder instability; Physical therapy

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial:
  Study intervention: apprehension-based training Control intervention: standard physical therapy
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Apprehension-based training (Experimental): Apprehension-based training is a 3-phase exercise intervention intended to expose patients to progressively increased shoulder apprehension-provoking conditions. Patients progress from one phase to the other upon completion of the previous level of exercise
  Interventions: Behavioral: Apprehension-based training
- Standard physical therapy (Active Comparator): Standard physical therapy will be provided by a licensed physical therapist and may include exercises of different kinds, manual therapy, dry needling or electrophysiological modalities.
  Interventions: Behavioral: Standard physical therapy

INTERVENTIONS:
Behavioral: Apprehension-based training — This intervention is comprised of the 3 phases:
  Static phase - Isometric (static) exercises performed in progressively greater shoulder apprehension ("instability") provoking conditions Dynamic phase: Isotonic (dynamic) exercises using shoulder apprehension-provoking movement patterns at a gradually increasing pace of movement.
  Neurocognitive phase: Dynamic phase exercises are continued at a high pace with the addition of cognitive tasks ("distractions").
  The intervention is guided by a physical therapist and includes up to 8 individual (one on one) sessions. In each session the physical therapist assesses exercise performance quality and when appropriate progresses exercise intensity and/or phase. Patients are expected to perform home exercises according to their phase of the program on a daily basis in between physical therapy sessions.
  Arms: Apprehension-based training
Behavioral: Standard physical therapy — Standard physical will be provided based on the assessment and judgment of the physical therapist. Intervention may include active exercises for increased shoulder mobility, muscle strength and neuromuscular control. Intervention may also include manual therapies such as massage, soft-tissue and joint mobilizations, dry needling, and electrophysiological modalities. No more than 8 individual sessions with a physical therapist will be provided over the course of treatment with some form of a home exercise program in between.
  Arms: Standard physical therapy

SUMMARY:
The goal of this clinical trial is to determine if a new rehabilitation protocol (apprehension-based training), leads to better recovery after shoulder dislocation among military personnel.

Participants will be randomly allocated to apprehension-based training or standard physical therapy. In apprehension-based training participants will train to control their shoulder under progressively more unstable conditions. Standard physical therapy will be provided based on the clinical judgment of the treating physical therapist The primary hypothesis is that participants undergoing apprehension-based training will experience a more complete recovery of function, better shoulder-related quality of life, and incur less recurrent dislocations.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-39 years
* Shoulder dislocation (primary or recurrent) documented by a medical practitioner (physician, military medic)
* Positive anterior apprehension test
* Gross shoulder muscle strength 3/5 or greater

Exclusion Criteria:

* Previous shoulder fracture, tendon tear, or shoulder surgery
* Voluntary shoulder dislocation
* Functional (Stanmore polar III) shoulder instability
* Dislocation associated with a motor vehicle accident.
* Diagnosis of rheumatoid arthritis, cancer (current), fibromyalgia, psychiatric disease)
* Current pregnancy
* Inability to attend at least one physical therapy session every 2 weeks.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 85 (Estimated)
Dates: Start 2025-02-05 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Return to preinjury level of function | 3 months following the end of intervention
  Patient's ability to resume their preinjury military and overall level of function will be assessed separately through a telephone interview 3 months after the end of their assigned intervention. This outcome will be rated dichotomously: "Yes" (have resumed my preinjury military/overall level of function), or "No" (have not been able to resume my preinjury military/overall level of function).
Western Ontario Shoulder Instability Index | Baseline to end of intervention (10 weeks) and 1-year follow-up (62 weeks).
  The Western Ontario Shoulder Instability Index is a self-reported measure of shoulder instability related quality of life. This questionnaire includes 21 items regarding symptoms, activity limitations, quality of life and emotions. Each item is scored on a 100mm visual analogue scale resulting in a total score of 0 - 2100 which can be converted to a percentage with greater scores indicating greater disability.
Recurrence | One year following the end of the intervention
  Recurrent events of instability, either in the form of a frank dislocation or a sensation of instability (subluxation) will be assessed through a telephone interview.
Supine moving apprehension test | Baseline to end of intervention (10 weeks)
  Dynamic stability will be assessed with the supine moving apprehension test. This is a functional performance test in which the patient is asked to repeatedly move the shoulder into 135- and 180-degrees of abduction from a supine position while holding a dumbbell (2-3 kg). The number of repetitions over one minute comprises the score of the test.

SECONDARY OUTCOMES:
Subjective shoulder value | Baseline, end of intervention (10 weeks), and 1-year follow up (62 weeks)
  A patient reported single numeric assessment of shoulder function as a percent of a normal shoulder: "What is the overall percent value of your shoulder if a completely normal shoulder represents 100%?"
Tampa scale of kinesiophobia | Baseline, end of intervention (10 weeks), and 1-year follow-up (62 weeks)
  A self-reported 17-item fear of movement and reinjury measure. Each item is scored on a 4-point Likert scale for a total score between 17-68.
Anterior apprehension test | Baseline to end of intervention (10 weeks)
  The sensation of apprehension will be assessed through the anterior apprehension test performed in 4 stages: 1.) shoulder abduction to 90 degrees; 2.) external rotation; 3.) horizontal abduction; 4.) Shoulder abduction beyond 90 degrees. Elicitation of apprehension (verbal, fascial expression, or muscle guarding) will be rated according to the stage at which it occurs (1-4). The test will be rated negative (5) if apprehension is not elicited at any stage.
Shoulder internal/external rotator muscle strength | Baseline and end of intervention (10 weeks)
  Shoulder internal and external rotator muscle strength will be assessed using a hand-held dynamometer in a supine-lying position with the shoulder abducted 90 degrees, neutral rotation, and the elbow bent 90 degrees. The examiner will position a hand-held dynamometer over the distal anterior (internal rotator strength) or posterior (external rotator strength) aspect of the forearm and resist a maximal voluntary effort by the patient. two repetitions will be performed for each strength test with the highest value used for data analysis.
Abdominal rollout | Baseline and end of intervention (10 weeks)
  From a kneeling position with the hands gripping a barbell loaded with a 5kg plate on each side, the patient will roll forward to the greatest distance possible and return to the starting position. The test will be performed in a narrow (shoulder width) and wide (2x shoulder width) hand grip. Up to 5 repetitions will be allowed to achieve maximum distance in each grip condition.
Heart rate variability | Baseline and end of intervention (10 weeks).
  Heart rate variability (HRV) during apprehension provocative and non-apprehension provocative shoulder movements will be measured using a Polar H10 chest strap. Heart rate variability will serve a physiological marker for autonomic nervous system response to movement provoked stress in the context of anterior shoulder dislocation.

CONTACTS AND LOCATIONS:
Overall Officials: Alon Rabin, PhD, DPT, Study Chair — Ariel University
Locations (1):
- Israel Defense Forces Medical Corps, Be’er Ya‘aqov, Israel

IPD SHARING:
Plan to Share IPD: Yes
Baseline, final and follow-up self-reported and physical performance outcome measures will be shared electronically.
Supporting Information: Study Protocol, SAP
Time Frame: 1.1.2028-1.1.2029
Access Criteria: Scholars, medical professionals as well as the general public may access outcomes measures data, intervention protocol and statistical analyses upon request from the principal investigator at the URL provided below.
URL: https://pniot.ariel.ac.il/projects/trp/GeneralInformation.asp?numRec=76&numtafrit=1&id_lang=1&d=

REFERENCES:
- [Background] Rabin A, Noyman L, Yaakobi N, Kazum E. Apprehension-Based Training: A Novel Treatment Concept for Anterior Shoulder Dislocation - A Case Report. Int J Sports Phys Ther. 2024 Jul 1;19(7):888-897. doi: 10.26603/001c.118928. eCollection 2024. PMID 38966825
- [Background] Rabin A, Chechik O, Olds MK, Uhl TL, Kazum E, Deutsch A, Citron E, Cohen T, Dolkart O, Bibas A, Maman E. The supine moving apprehension test-Reliability and validity among healthy individuals and patients with anterior shoulder instability. Shoulder Elbow. 2024 Feb;16(1):98-105. doi: 10.1177/17585732231170197. Epub 2023 Apr 18. PMID 38435037